CLINICAL TRIAL: NCT06785779
Title: Survey Assessing Prospective Patient's Short-term Treatment Satisfaction and Quality of Life in Patients With Hidradenitis Suppurativa Initiated on Cosentyx (Secukinumab) in Routine Clinical Practice in Saudi Arabia: ILLUMINATE-SA
Brief Title: Short-term Treatment Satisfaction in Hidradenitis Suppurativa Patients Initiated on Cosentyx in Routine Clinical Practice in Saudi Arabia
Acronym: ILLUMINATE-SA
Status: Recruiting | Type: Observational
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Other Study IDs: CAIN457MSA01
Record Dates: First submitted 2025-01-13; First posted 2025-01-21 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Hidradenitis Suppurativa (HS)
Keywords: Hidradenitis Suppurativa; HS; secukinumab; NIS; Saudi Arabia
MeSH Terms: conditions — Hidradenitis Suppurativa | interventions — secukinumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Secukinumab: Patients who are newly initiated on Secukinumab
  Interventions: Other: Secukinmab

INTERVENTIONS:
Other: Secukinmab — This is an observational study. There is no treatment allocation. The decision to initiate secukinumab will be based solely on clinical judgement.
  Other Names: Cosentyx

SUMMARY:
This study aims to assess the treatment satisfaction of HS patients newly started on secukinumab in Saudi Arabia, in terms of patient reported convenience, perceived safety, perceived effectiveness and global treatment satisfaction as measured by the treatment satisfaction questionnaire for medication (TSQM) at week 24 among moderate to severe HS patients.

DETAILED DESCRIPTION:
This is a 24-week longitudinal single arm prospective study based on data collected from electronic medical records (EMRs) and patient-reported outcomes questionnaires (TSQM, DLQI, and NPRS-11) to evaluate patient-reported satisfaction and early QoL experiences among HS adult patients who are newly administering Secukinumab as per routine clinical practice.

Data will be captured from both data sources (EMRs and Questionnaires) at the following time points (+/- 1 month):

* Baseline (index date: initiation of Secukinumab),
* 24 weeks.

This is in line with the frequency of routine follow-up visits and as per the standard of care to report on pre-defined outcomes in a representative HS population across Saudi Arabia.

ELIGIBILITY:
Inclusion Criteria:

1. Male or Female adult patients ≥18 years of age at the time of data collection.
2. Patient with a confirmed diagnosis of active moderate to severe HS.
3. Secukinumab naive patients (first dose to coincide within one month of the signature of the informed consent) as per locally approved label.
4. Patients can be using antibiotics or have undergone surgery as per routine clinical practice.
5. Patients agree to sign an informed consent form (ICF) to be able to complete the questionnaires.

Exclusion Criteria:

1. Patients not fulfilling any of the above-mentioned inclusion criteria.
2. Patient's refusal to be included in the study or refusal to sign the ICF.
3. A history of off-label indication uses of biological treatment or JAK inhibitor.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who are newly initiated on Secukinumab as per locally approved labels and routine clinical practice will be enrolled over a period of 6 months and followed up for 24 weeks to assess study outcomes
Sampling Method: Non-Probability Sample
Enrollment: 77 (Estimated)
Dates: Start 2025-03-10 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Mean Score in the Treatment Satisfaction Questionnaire (TSQM) | Week 24
  TSQM questionnaire consists of 14 questions with a score ranging from 0 to 100. The questionnaire has four subscales, effectiveness (3 questions), side Effects (5 questions), convenience (3 questions) and global Satisfaction (3 questions).
  TSQM scoring is calculated by each subscale, which ranges from 0 to 100, with higher scores indicating higher patient satisfaction with medication.

SECONDARY OUTCOMES:
Mean change from baseline in patient-reported QoL via the Dermatology Life Quality Index (DLQI) Questionnaire | Baseline, week 24
  The DLQI is a valid 10-item instrument used to measure the impact of skin diseases on a patient's quality of life. Each question is scored on a scale of 0 to 3, with 0 indicating "not at all" and 3 indicating "very much." The total score ranges from 0 to 30, with a higher score indicating a greater impact on the patient's quality of life.
Mean change from baseline to week 24 in the Numeric Pain Rating Scale (NPRS-11) | Baseline, week 24
  NPRS-11 is a subjective measure representing pain intensity in which individuals rate their pain on an eleven-point numerical scale. The scale is composed of 0 (no pain at all) to 10 (worst imaginable pain)
Baseline characteristics-age | Baseline
  Age at baseline (years)
Baseline characteristics - Ethnicity | Baseline
  Assessment of Participant's ethnicity
Baseline characteristics - Socio-economic status | Baseline
  Assessment of socio-economic status
Baseline characteristics - smoking status | Baseline
  Assessment of smoking status
Baseline characteristics - Family history of HS | Baseline
  Number of participants with family history of HS
Baseline characteristics - Duration of the disease | Baseline
  Time since- symptom onset and/or diagnosis
Baseline characteristics - Previous HS-related treatment | Baseline
  Number of participants with Previous HS- related treatment including treatment type
Baseline characteristics - previous HS-related surgeries | Baseline
  Number of participants with Previous HS- related surgeries including surgery type
Baseline characteristics - Current or previous use of antibiotic treatment | Baseline
  Number of participants with current or previous use of antibiotic treatment including antibiotic type.
Baseline characteristics - Time since diagnosis to first treatment and secukinumab treatment | Baseline
  Time from diagnosis to start the first treatment and Time from diagnosis to start of Secukinumab
Baseline characteristics - concomitant medications | Baseline
  Assessment of concomitant medications
Baseline characteristics - Hurley Stage | Baseline
  Classification of HS severity assessed by Hurley staging scale, Stage I (Mild) , Stage II (Moderate) and stage III (Severe)
Baseline characteristics - number of inflammatory nodules, abscesses and draining tunnels/fistula | Baseline
  Number of inflammatory nodules, abscesses and draining tunnels/fistula

CONTACTS AND LOCATIONS:
Locations (3):
- Saudi Arabia (3):
  - Novartis Investigative Site, Riyadh, SAU
  - Novartis Investigative Site, Jeddah
  - Novartis Investigative Site, Riyadh

IPD SHARING:
Plan to Share IPD: No